CLINICAL TRIAL: NCT01703767
Title: Gulf War 1 Veteran Patient Satisfaction With VA Primary Care: A Survey Study.
Brief Title: Gulf War 1 Veteran Healthcare Satisfaction
Status: Withdrawn | Type: Observational
Why Stopped: We did not have sufficient funds to conduct the study.
Sponsor: University of Utah (Other)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Gavin West, Associate Chief of Medicine, VASLCHCS, University of Utah
Other Study IDs: IRB_00053707
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Persian Gulf War Syndrome in Veteran
Keywords: patient satisfaction; Gulf War 1 Veteran; Desert Storm Veteran
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gulf War 1 Veterans: Persian Gulf War 1 Veterans (GW1V) who are currently treated by a primary care physician at the VA Salt Lake City Health Care System. GW1V will assess their primary care satisfaction before and after their providers receive a Provider Education Workshop.
  Interventions: Behavioral: Provider Education Workshop

INTERVENTIONS:
Behavioral: Provider Education Workshop — Educational resources for physicians regarding the needs of GW1V patients.

SUMMARY:
The purpose of this study is to investigate Gulf War 1 Veteran (GW1V) patient perceptions of, and satisfaction with, their VA primary care treatment, and physician effectiveness in delivering improved point of service, in the Primary Care Clinics at the Veterans Administration (VA) Salt Lake City Health Care System.

DETAILED DESCRIPTION:
Veterans of the 1990-1991 Gulf War1 (GW1) conflict are still experiencing a host of adverse health conditions at the present time. Many GW1 Veterans are still unhappy with their health care at the VA, and other stakeholders are critical of how the VA has dealt with GW1 Veterans' issues. For these reasons, the Gulf War Veterans' Illness Task Force (GWVI-TF) was set up to find ways to improve the situation.

The present survey study addresses one of GWVI-TF's missions, that is, to identify gaps in VA services, and to discover opportunities to better serve GW1V. Caring for GW1V is a top priority for VA health care providers, which is all the more pressing for the following reasons: 1. medical science of Gulf War Illness and environmental exposures is still at its infancy, 2. most providers have not received any focused education about how to take care of GW1V and the unique medical problems these veterans face, 3. a lack of provider knowledge that GW1V may receive may lead to decreased satisfaction on the part of GW1V and may result in GW1V perceived health service quality that is compromised.

In this pilot study, we focus on #2 and #3, to determine how we may understand veterans' perceptions of their medical treatment to ultimately improve GW1V medical health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a gulf war Veteran who served during the Persian Gulf War (GW1) of 1990-1991
* currently treated by a primary care physician at the VASLCHCS

Exclusion Criteria:

* cannot read and write English

Ages: 38 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persian Gulf War Veterans who are currently treated by a primary care physician at the VASLCHCS Blue Clinic and West Valley Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Change in Client Satisfaction score | baseline and 3 months
  The Client Satisfaction Questionnaire will be used to measure change in client satisfaction at baseline and after providers have received Provider Education Workshop training
Change in Patient Satisfaction score | baseline and 3 months
  The Patient Satisfaction Questionnaire will be used to measure change in patient satisfaction at baseline and after providers have received Provider Education Workshop training

SECONDARY OUTCOMES:
Change in Physician Assessment of GW1V Care | Baseline and 3 months
  The Physician Survey will be used to measure change in physician assessment of GW1V care at baseline and after providers have received Provider Education Workshop training.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin West, MD, Principal Investigator — VA Salt Lake City Health Care System
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - VA SLC Health Care System, Salt Lake City, Utah